CLINICAL TRIAL: NCT06125678
Title: Correlation and Assessment of Small Bowel Lesion Using Cross Sectional Imaging Techniques Compared to Small Intestinal Contrast Ultrasonography in Known Small Bowel Crohn's Disease(the CACTUS-CD Trial): a Prospective Study
Brief Title: Correlation of Cross Sectional Imaging and Small Intestinal Contrast Ultrasonography in Known Crohn's Disease
Acronym: CACTUS-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AIG/IEC-BH&R 49 / 06.2023-04
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease; Ultrasound Therapy; Complications; Computed Tomography; Magnetic Resonance Imaging
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Small intestinal contrast enhanced ultrasound followed by cross sectional imaging (Experimental): Patients shall be undergoing small intestinal contrast enhanced ultrasound followed by cross sectional imaging
  Interventions: Diagnostic Test: Small intestinal contrast enhanced ultrasound followed by Computed tomography/Magnetic resonance enterography

INTERVENTIONS:
Diagnostic Test: Small intestinal contrast enhanced ultrasound followed by Computed tomography/Magnetic resonance enterography — First small intestinal contrast enhanced ultrasound shall be done followed by CT enterography or MR enterography

SUMMARY:
Small intestinal contrast ultrasound (SICUS) is a modality of intestinal ultrasound (IUS) which does not require any parenteral administration of contrast agent but requires ingestion of around 500 ml of polyethylene glycol (PEG). SICUS does not involve any radiation. Computed tomography enteroclysis (CTE) requires colonic cleansing using polyethylene glycol (PEG) followed by infusion of 1.5 litres of PEG via a nasal catheter to distend and properly visualise the small intestine. CTE although accurate for assessing response to therapy and transmural healing in small bowel CD is associated with radiation and adds to cost of management. Magnetic resonance enterography (MRE) using PEG followed by 2 liters of oral fluid with mannitol was administered to distend and properly visualize the small intestine. MRE although accurate for assessing response to therapy and transmural healing in small bowel CD is associated with radiation and adds to cost of management. On the other hand, SICUS is relatively non-invasive method of small bowel assessment although the accuracy has not been studied prospectively. An earlier retrospective study in which MRE/CTE and SICUS are done within 3 months of each other, SICUS had identified lesions and complications in patients with CD with high levels of sensitivity, specificity, and accuracy compared to CT-enteroclysis (3). These findings need prospective validation. The accuracy of SICUS may be suboptimal due to constant peristalsis in the small intestine. Hence the investigators planned this study to perform SICUS in patients with small bowel CD who otherwise require a MRE/CTE for disease monitoring on the same day before the procedure with the same PEG preparation. If SICUS findings are found to correlate with MRE/CTE findings intros study, SICUS have the potential to replace other modalities for monitoring of small bowel Crohn's disease (CD) and emerge as a cost-effective, easy alternative. The investigators also want to understand the drawbacks and limitations of SICUS in this scenario.

DETAILED DESCRIPTION:
Diagnosis, CD site and patient's management shall be made according generally accepted recommendations(4). SICUS shall be performed in all participants by one independent experienced operator (MAM). Colonic cleansing shall be done on night before the examination with Polyethylene glycol (PEG) solution (1 litre). The participants shall be examined after the ingestion of 375 mL (range 250-500 mL) of polyethylene glycol (PEG) in the morning using a convex transducer (2-6 MHz) and a high frequency linear-array transducer for details (5-14 MHz). Median SICUS duration shall be noted. SICUS shall be performed without any additional charges to the participant. CT-Enteroclysis shall be performed in all participants by one independent experienced operator (UK). A 20G needle shall be placed in an antecubital vein and 8-F nasojejunal catheter with aTeflon-covered guide wire shall be positioned under fluoroscopic guidance with the distal extremely located in the distal duodenum/proximal jejunum. Afterward the patient shall be taken into the CT room where hypodense contrast material (1500 mL of PEG) shall be administered manually with 60-mL syringes, with a constant and continuous injection rate of 150 mL/min followed by a flow rate of 200 mL/min until the maximum tolerance of the patient. Just before the examination participants shall receive a smooth muscle relaxant (N butyl 4 scopolamine) to prevent spasms, achieve uniform small bowel distension, and reduce abdominal discomfort. The study shall be performed by a 64-slice multidetector CT with the following scan parameters: collimation 1.25 mm, table feed 39.37 mm/rot, 120 kV, 300 mAs,pitch 0.984:1, rotation time 0.5 s, time of acquisition 12.5 s, FOV 50 cm, matrix 512x512. After the infusion of PEG, CT scan seal be performed before and after the administration of intravenous iodinated contrast material. The contrast-enhanced study shall be acquired 70s after the administration of contrast material (Ultravist 370, Schering AG, Berlin, Germany). Median CT-Enteroclysis duration shall be recorded. Magnetic Resonance enterography (MRE) shall be performed in all participants by one independent experienced operator. The participant shall be fasted for 4-6 h prior to the study. In adults, 2 liters of oral fluid with mannitol shall be administered to distend the bowel loops. Just before the examination participants shall receive a smooth muscle relaxant (Buscopan) to prevent spasms, achieve uniform small bowel distension, and reduce abdominal discomfort. T2, BTFE(axial and coronal sequence),diffusion weighted imaging (DWI)(Coronal sequence), Post contrast (Axial, Coronals and sagittal sequence) will be taken.Median MRE duration shall be recorded.The site of small bowel involvement, maximal bowel wall thickness and complications like stricture and fistula detected by SICUS and MRE/CTE shall be collected and correlated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known small bowel CD beyond reach of standard endoscopy who warrants monitoring of disease status either due to assessment of response to therapy/relapse/new unexplained symptoms, persistent disease activity, prior to switching therapy or deciding on surgical management.

Exclusion Criteria:

* Obese patients with poor ultrasound window
* pregnant/lactating mother
* Not willing for CT or enteroclysis examination
* Renal insufficiency precluding CT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Change in management decision after cross sectional imaging compared to ultrasound | Day 1
  Percentage of patients in which cross sectional imaging changed the management decision

SECONDARY OUTCOMES:
Correlation between bowel wall thickness in affected area in small intestine between small intestinal contrast ultasonography and cross sectional imaging | Day 1
  Correlation between bowel wall thickness in ultrasonography and cross sectional imaging based on correlation coefficient
Agreement for extent of involvement in affected area of small intestine between small intestinal contrast ultasound and cross sectional imaging | Day 1
  Percentage of patients in which small intestinal ultrasound correctly identified extent of involvement compared to cross sectional imaging
Agreement for detecting complications between small intestinal contrast ultrasound and cross sectional imaging | Day 1
  Percentage of patients in which small intestinal ultrasound correctly identified complications compared to cross sectional imaging

CONTACTS AND LOCATIONS:
Overall Officials: Partha Pal, MD, DrNB, Principal Investigator — Asian Institute of Gastroenterology and Asian Healthcare Foundation
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pal P, Mateen MA, Pooja K, Marri UK, Reddy CR, Salman S, Piprikar R, Gupta R, Tandan M, Reddy DN. Correlation and Assessment of Small Bowel Lesions Using Cross-Sectional Imaging Techniques Compared With Small Intestinal Contrast Ultrasonography in Known Crohn's Disease (the CACTUS-CD Study): A Paired, Prospective, Confirmatory Study. Am J Gastroenterol. 2025 Sep 29. doi: 10.14309/ajg.0000000000003776. Online ahead of print. PMID 41020653